CLINICAL TRIAL: NCT03358784
Title: A Multi-center Study on Comparison of Hemi-shoulder Arthroplasty and PHILOS in Treating Three or Four-part Fractures of Proximal Humerus.
Brief Title: Comparison of Hemi-shoulder Arthroplasty and PHILOS in Treating Three or Four-part Fractures of Proximal Humerus
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Zhang Peixun, Department of orthopaedics and trauma, Peking University People's Hospital
Other Study IDs: PUPH2017PHF
Record Dates: First submitted 2017-11-26; First posted 2017-12-02 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Humeral Fracture, Proximal
Keywords: Humeral Fractures, Proximal; Arthroplasty, Shoulder Replacement; Bone Plates
MeSH Terms: conditions — Shoulder Fractures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PHILOS Plate: three or four-part fractures of proximal humerus treated with internal fixation
  Interventions: Procedure: PHILOS Plate
- Hemi-shoulder arthroplasty: three or four-part fractures of proximal humerus treated with hemi-shoulder arthroplasty
  Interventions: Procedure: Hemi-shoulder Arthroplasty

INTERVENTIONS:
Procedure: Hemi-shoulder Arthroplasty — Hemi-shoulder Arthroplasty treating three or four-part fractures of proximal humerus
  Groups: Hemi-shoulder arthroplasty
Procedure: PHILOS Plate — PHILOS plate treating three or four-part fractures of proximal humerus
  Groups: PHILOS Plate

SUMMARY:
To explore clinical effectiveness of PHILOS plate fixation and hemi-shoulder arthroplasty in treating three or four-part fractures of proximal humerus

DETAILED DESCRIPTION:
From April 2015 and April 2017, patients from multi-center aged over 60 years old with three and four-part fractures of proximal humerus were treated with Proximal Humerus Internal Locking System(PHILOS) and hemi-shoulder arthroplasty in multi-center. All the patients received the same rehabilitation course. At 6 months after surgery, postoperative complications were observed, EQ-5D was used to evaluate quality of life, and ASES score was used to assess functional outcomes.

ELIGIBILITY:
Inclusion Criteria:

three or four part fractures of proximal humerus

Exclusion Criteria:

1. Severe comminuted fractures of proximal humerus
2. past history of injured-side shoulder surgery
3. Patients who cannot tolerate surgery

Ages: 60 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with three or four part fractures of proximal humerus, who agreed to receive surgery.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-03-05 (Estimated); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications | 6 months after surgery
  Postoperative complications were observed

SECONDARY OUTCOMES:
EQ-5D | 6 months after surgery
  EQ-5D was used to evaluate quality of life
ASES score | 6 months after surgery
  ASES was used to assess functional outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Peixun Zhang, MD, Principal Investigator — Peking University People's Hospital

IPD SHARING:
Plan to Share IPD: No